CLINICAL TRIAL: NCT04459741
Title: Hypertension, Dietary Salt and Inflammation
Brief Title: HIV, Immune Activation and Salt Sensitive Hypertension
Acronym: HISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mulungushi University (Other)
Collaborators: University of Zambia (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sepiso K. Masenga, Dr, Mulungushi University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: SKM001
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: HIV-1-infection; Hypertension,Essential
Keywords: Inflammation; Human immunodeficiency virus (HIV); Salt; Interleukin 6; Interleukin 17A; Hypertension
MeSH Terms: conditions — Essential Hypertension; Inflammation; Acquired Immunodeficiency Syndrome; Hypertension | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants are instructed on salt deprivation for a week followed by a low salt (4 grams) diet for one week and switched to high salt (9 grams) for the following one week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIV+ Hypertensive (Experimental): Participants receive 4 grams of dietary salt (equivalent of 1, 560 mg sodium) everyday for seven days followed by 9 grams (equivalent of 3, 510 mg sodium) of dietary salt for the following seven days
  Interventions: Dietary Supplement: Dietary salt (Sodium chloride)
- HIV+ Normotensive (Other): Participants receive 4 grams of dietary salt (equivalent of 1, 560 mg sodium) everyday for seven days followed by 9 grams (equivalent of 3, 510 mg sodium) of dietary salt for the following seven days
  Interventions: Dietary Supplement: Dietary salt (Sodium chloride)
- HIV- Hypertensive (Experimental): Participants receive 4 grams of dietary salt (equivalent of 1, 560 mg sodium) everyday for seven days followed by 9 grams (equivalent of 3, 510 mg sodium) of dietary salt for the following seven days
  Interventions: Dietary Supplement: Dietary salt (Sodium chloride)
- HIV- Normotensive (Other): Participants receive 4 grams of dietary salt (equivalent of 1, 560 mg sodium) everyday for seven days followed by 9 grams (equivalent of 3, 510 mg sodium) of dietary salt for the following seven days
  Interventions: Dietary Supplement: Dietary salt (Sodium chloride)

INTERVENTIONS:
Dietary Supplement: Dietary salt (Sodium chloride) — Dietary salt used was sodium chloride tablets (from the research consolidated midland corporation division, New York, USA) which participants crashed and put in their food and/or ingested. Each tablet weighed one (1) gram and contained 394 mg of sodium and 606 mg of chloride.

SUMMARY:
High dietary salt is associated with immune activation, elevated levels of inflammatory cytokines and hypertension in murine models. Hypertension is independently associated with inflammation in both murine studies and studies in humans. In people living with HIV, these interactions are not well established. The aim of this study is to determine the effect of excess dietary salt on immune cell activation, pro- and anti-inflammatory cytokines and blood pressure between individuals with and without hypertension among people living with HIV and HIV negative persons.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 and above) who will be required to verbally consent and sign a consent form
* HIV positive or HIV Normotensive individuals or hypertensive If HIV, on antiretroviral therapy ART treated hypertensive individuals

Exclusion Criteria:

* Existence of comorbidities such as diabetes mellitus and cancer Existing and recent past opportunistic infections, syphilis, hepatitis C and B virus infection and tuberculosis infection;
* Sick persons (clients seeking healthcare due to an illness rather than routine ART clinic reviews)
* Those with recent and current alcohol consumption and smoking status

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Pro-inflammatory cytokines | 2 weeks: At the end of the low- and high-salt phases
  Elevated levels of pro-inflammatory cytokines when compared between low and high salt phase

SECONDARY OUTCOMES:
Blood pressure | 2 weeks: At the end of the low- and high-salt phases
  Elevated blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Sepiso K Masenga, PhD, Principal Investigator — Mulungushi University
Locations (1):
- Livingstone Central Hospital, Livingstone, Southern Province, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masenga SK, Hamooya BM, Nzala S, Kwenda G, Heimburger DC, Mutale W, Koethe JR, Kirabo A, Munsaka SM. HIV, immune activation and salt-sensitive hypertension (HISH): a research proposal. BMC Res Notes. 2019 Jul 16;12(1):424. doi: 10.1186/s13104-019-4470-2. PMID 31311574